CLINICAL TRIAL: NCT05839327
Title: Impact of Mental Health and Cognitive Disorders on Quality of Life in Severe Covid-19
Brief Title: Impact of Mental Health and Cognitive Disorders on Quality of Life in Severe Covid-19 Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, ICU Assistent Physician, Hospital Sao Domingos
Other Study IDs: 15/2023
Record Dates: First submitted 2023-04-30; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Post-Intensive Care Syndrome
Keywords: COVID-19; Critically ill patients; Cognitive disorders; Post-traumatic stress disorder; Anxiety; Depression; Post-intensive care syndrome
MeSH Terms: conditions — COVID-19 post-intensive care syndrome; COVID-19; Cognitive Dysfunction; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Montreal cognitive assessment scale (MOCA) — Tests to evaluate cognitive disorders (MOCA), anxiety and depression (HADS) Pos-traumatic stress disorder (PCL-C) and quality of life (SF-36)
  Other Names: Hospital anxiety and depression scale ( HADS); Post-traumatic stress disorder checklist civilian version (PCL-C); Short form health survey 36 (SF-36)

SUMMARY:
The objective of this single-center retrospective observational study is to describe cognitive and psychological outcomes and their impact on quality of life after at least 3 months of intensive care unit (ICU) discharge in severe COVID-19 survivors.

DETAILED DESCRIPTION:
Background: The COVID-19 pandemic has already affected more than 600 million people worldwide and resulted in at least 6 million deaths (https:coronavirus.jhu.edu/map.html). The pandemic has also resulted in a growing population of individuals recovering from acute SARS-CoV-2 infection. Accumulating observational data suggest that these patients often experience a wide range of symptoms after recovery from acute illness. The dysfunctions ranging from motor, cognitive disability, anxiety, depression and post-traumatic stress disorder. However, there is still unknown data about the occurrence of mental health manifestations after a critical illness and their consequences in mid term quality of life.

Purpose: Many patients with coronavirus disease 2019 (COVID-19) required critical care. Mid-term outcomes of the survivors need to be assessed. The objective of this single-center retrospective observational study is to describe their cognitive and psychological outcomes and their impact on quality of life afer at least 3 months following intensive care unit (ICU)-discharge.

Objectives: Our objective will be to evaluate the incidence of non-physical post-intensive care syndrome, such as symptoms of anxiety, depression, cognitive and post-traumatic stress disorder (PTSD) after hospital discharge in our severe COVID-19 population, as well as determining their long-term consequences in quality of life (QoL).

Methods: An observational retrospective study will be conducted, including all patients with severe COVID-19 admitted to the intensive care unit of a private tertiary hospital from April 2020 to October 2021. Patients were routinely assessed after 3 months of ICU discharge in our multidisciplinary follow-up clinic. A trained research team routinely applied the Montreal Cognitive Assessment Scale (MOCA), Hospital Anxiety and Depression Scale (HADS), PCL-C (Post-traumatic Stress Disorder Checklist: Civilian Version) and Short Form Health Survey 36 (SF-36), during the follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All 18 years and older patients with severe COVID-19, confirmed by real-time reverse transcriptase-polymerase chain reaction., admitted to a 15- bed intensive care unit of a tertiary hospital from April 2020 to October 2021.

Exclusion Criteria:

* Still hospitalized or inpatient in rehabilitation facility
* Previous cognitive impairmant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with coronavirus disease 2019 (COVID-19) admitted to intensive care unit requiring invasive and non-invasive respiratory support evaluated at least 3 months after hospital discharge for cognitive and psycological components of post-intensive care syndrome and the impact on quality of life.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-02-10 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale (MOCA) | 6 months after hospital discharge
  The MoCA total score was used for analysis: it ranges from 0 to 30, the lower scores indicating worse cognitive performances. The validated cut-off of 26 was used to distinguish light cognitive disorders (≥ 26) and proven cognitive impairments (< 26)
  The MoCA total score was used for analysis: it ranges from 0 to 30, the lower scores indicating worse cognitive performances. The validated cut-off of 26 was used to distinguish light cognitive disorders (≥ 26) and proven cognitive impairments (< 26)
  The MoCA total score was used for analysis: it ranges from 0 to 30, the lower scores indicating worse cognitive performances. The validated cut-off of 26 was used to distinguish light cognitive disorders (≥ 26) and proven cognitive impairments (< 26)
  The MOCA total score was used for analysis: it ranges from 0 to 30, the lower scores indicating worse cognitive performances. The validated cut-off of 26 was used to distinguish light cognitive disorder (> 26) and
Hospital Anxiety and depression scale (HADS) | 6 months after hospital discharge
  The HADS consists of two 7-item subscales evaluating symptoms of depression (seven items-HADS-D subscale) and symptoms of anxiety (seven items-HADS-A subscale). The standard cutoff threshold value of > 7 out of 21 on either subscale was used to define a borderline status (score 8 to 10) or clinically significant status (score 11 to 21) of depression or anxiety, respectively.
Post-traumatic Stress Disorder Checklist: Civilian Version (PCL-C) | 6 months after hospital discharge
  PCL-C is an instrument designed to assess the consequences of a number of different types of traumatic experience. To complete the questionnaire, the subject should gauge to what extent they have been disturbed by the symptoms described during the previous month, using a scale of severity from 1 to 5 (not at all to very much). It defines a score greater than or equal to 3 (average) for any of the 17 items as clinically significant.
  PCL-C is an instrument designed to assess the consequences of a number of different types of traumatic experience. To complete the questionnaire, the subject should gauge to what extent they have been disturbed by the symptoms described during the previous month, using a scale of severity from 1 to 5 (not at all to very much). It defines a score greater than or equal to 3 (average) for any of the 17 items as clinically significant.

SECONDARY OUTCOMES:
Mental Component Summary (MCS) of Short Form- 36 (SF-36) Instrument | 6 months after hospital discharge
  MCS is composed of scales assessing mental function, role limitations caused by mental problems, bodily pain and general health. The result scale ranges from 0 to 100, with 0 being the worst result and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: JOAQUIM C LOBATO FILHO, MD, Principal Investigator — Hospital Sao Domingos; JOSE R AZEVEDO, MD, PhD, Study Chair — Hospital Sao Domingos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambermont B, Rousseau AF, Seidel L, Thys M, Cavalleri J, Delanaye P, Chase JG, Gillet P, Misset B. Outcome Improvement Between the First Two Waves of the Coronavirus Disease 2019 Pandemic in a Single Tertiary-Care Hospital in Belgium. Crit Care Explor. 2021 May 19;3(5):e0438. doi: 10.1097/CCE.0000000000000438. eCollection 2021 May. PMID 34079951
- [Result] Needham DM, Davidson J, Cohen H, Hopkins RO, Weinert C, Wunsch H, Zawistowski C, Bemis-Dougherty A, Berney SC, Bienvenu OJ, Brady SL, Brodsky MB, Denehy L, Elliott D, Flatley C, Harabin AL, Jones C, Louis D, Meltzer W, Muldoon SR, Palmer JB, Perme C, Robinson M, Schmidt DM, Scruth E, Spill GR, Storey CP, Render M, Votto J, Harvey MA. Improving long-term outcomes after discharge from intensive care unit: report from a stakeholders' conference. Crit Care Med. 2012 Feb;40(2):502-9. doi: 10.1097/CCM.0b013e318232da75. PMID 21946660
- [Result] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Result] Martillo MA, Dangayach NS, Tabacof L, Spielman LA, Dams-O'Connor K, Chan CC, Kohli-Seth R, Cortes M, Escalon MX. Postintensive Care Syndrome in Survivors of Critical Illness Related to Coronavirus Disease 2019: Cohort Study From a New York City Critical Care Recovery Clinic. Crit Care Med. 2021 Sep 1;49(9):1427-1438. doi: 10.1097/CCM.0000000000005014. PMID 33769771
- [Result] Mongodi S, Salve G, Tavazzi G, Politi P, Mojoli F; COVID-19 Post-ICU team; COVID-19 Pavia Crisis Unit. High prevalence of acute stress disorder and persisting symptoms in ICU survivors after COVID-19. Intensive Care Med. 2021 May;47(5):616-618. doi: 10.1007/s00134-021-06349-7. Epub 2021 Mar 17. No abstract available. PMID 33730197
- [Result] Ramani C, Davis EM, Kim JS, Provencio JJ, Enfield KB, Kadl A. Post-ICU COVID-19 Outcomes: A Case Series. Chest. 2021 Jan;159(1):215-218. doi: 10.1016/j.chest.2020.08.2056. Epub 2020 Aug 21. No abstract available. PMID 32835708
- [Result] Valent A, Dudoignon E, Ressaire Q, Depret F, Plaud B. Three-month quality of life in survivors of ARDS due to COVID-19: A preliminary report from a French academic centre. Anaesth Crit Care Pain Med. 2020 Dec;39(6):740-741. doi: 10.1016/j.accpm.2020.10.001. Epub 2020 Oct 10. No abstract available. PMID 33049394
- [Result] Writing Committee for the COMEBAC Study Group; Morin L, Savale L, Pham T, Colle R, Figueiredo S, Harrois A, Gasnier M, Lecoq AL, Meyrignac O, Noel N, Baudry E, Bellin MF, Beurnier A, Choucha W, Corruble E, Dortet L, Hardy-Leger I, Radiguer F, Sportouch S, Verny C, Wyplosz B, Zaidan M, Becquemont L, Montani D, Monnet X. Four-Month Clinical Status of a Cohort of Patients After Hospitalization for COVID-19. JAMA. 2021 Apr 20;325(15):1525-1534. doi: 10.1001/jama.2021.3331. PMID 33729425
- [Result] McCue C, Cowan R, Quasim T, Puxty K, McPeake J. Long term outcomes of critically ill COVID-19 pneumonia patients: early learning. Intensive Care Med. 2021 Feb;47(2):240-241. doi: 10.1007/s00134-020-06313-x. Epub 2020 Nov 9. No abstract available. PMID 33169214
- [Result] Huang C, Huang L, Wang Y, Li X, Ren L, Gu X, Kang L, Guo L, Liu M, Zhou X, Luo J, Huang Z, Tu S, Zhao Y, Chen L, Xu D, Li Y, Li C, Peng L, Li Y, Xie W, Cui D, Shang L, Fan G, Xu J, Wang G, Wang Y, Zhong J, Wang C, Wang J, Zhang D, Cao B. 6-month consequences of COVID-19 in patients discharged from hospital: a cohort study. Lancet. 2021 Jan 16;397(10270):220-232. doi: 10.1016/S0140-6736(20)32656-8. Epub 2021 Jan 8. PMID 33428867
- [Result] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Jenkinson C, Layte R, Jenkinson D, Lawrence K, Petersen S, Paice C, Stradling J. A shorter form health survey: can the SF-12 replicate results from the SF-36 in longitudinal studies? J Public Health Med. 1997 Jun;19(2):179-86. doi: 10.1093/oxfordjournals.pubmed.a024606. PMID 9243433